CLINICAL TRIAL: NCT02004483
Title: Comprehensive Analysis of Myocardial Layer Specific Systolic and Diastolic Function in Patients With Coronary Artery Disease Undergoing Percutaneous Coronary Intervention
Brief Title: Analysis of Myocardial Layer Specific Systolic and Diastolic Function During and After PCI
Acronym: PCI-Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Department of Biomedical Engineering, Technion, Haifa, Israel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-091; 032/10 (Other: Ethics)
Record Dates: First submitted 2013-11-11; First posted 2013-12-09 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Percutaneous Coronary Intervention; Myocardial Ischemia; Anginal Pain
Keywords: percutaneous coronary intervention; ischemia; strain; coronary stenosis
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Ischemia; Sprains and Strains; Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Percutaneous Coronary Intervention (Experimental): Each patient will get elective percutaneous coronary angioplasty with balloon inflation(PCI). During and after PCI 2D-echography (strain) will be performed.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous coronary intervention is performed according to standard practice. Direct stenting is required for the procedure as it is done in most coronary interventions today. After insertion of the non-inflated stent into the coronary lesion there should still be flow to the distal vessel. The stent should be implanted at high-pressure with balloon inflation lasting for 60 seconds to allow adequate expansion of the stent. Post-dilatation should be performed if required. However, this should be done more than 5 minutes after stent implantation.

SUMMARY:
Investigators will analyzed systolic and diastolic function during and after ischemia induced by percutaneous coronary intervention.Also will be analyzed a local work index during acute ischemia induced by percutaneous coronary intervention.

DETAILED DESCRIPTION:
PART 1: ANALYSIS OF LAYER SPECIFIC SYSTOLIC AND DIASTOLIC FUNCTION DURING ACUTE ISCHEMIA INDUCED BY PERCUTANEOUS CORONARY INTERVENTION 35 patients with normal systolic left ventricular function at baseline with indication for elective percutaneous coronary angioplasty will be included in the study. In these patients acute ischemia will be induced by elective percutaneous coronary angioplasty with balloon inflation and thus vessel occlusion for 60 sec. During these 60 seconds ischemia will develop throughout all layers of the myocardium affecting diastolic systolic and diastolic function. During the subsequent reperfusion period signs of ischemia with systolic and diastolic dysfunction of all layers will subside. Echocardiographic imaging at short intervals of 10 sec during ischemia and at intervals of 20 sec during reperfusion up to 10 min after reopening of the vessel as well as 1 hour and 24 hours later will allow serial comparison of strain curves and thereby allow definition of the time sequence systolic and diastolic function abnormalities occur in three myocardial layers as well as the resolution of abnormalities during reperfusion. The analysis of circumferential as well as radial strain will allow definition of differences between radial and circumferential strain during ischemia induction and resolution.

PART 2: ANALYSIS OF LOCAL WORK INDEX DURING ACUTE ISCHEMIA INDUCED BY PERCUTANEOUS CORONARY INTERVENTION.

In the same 35 patients as in Clinical step 1 the local work index of the ischemic area as well as the contralateral non-ischemic areas will be determined in serial studies to determine the onset of abnormality, the amount of abnormality and the resolution of abnormality. Changes in local work index in the ischemic area will be related to changes in peak systolic strain and strain imaging diastolic index.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Adequate quality of echocardiographic images.
* Significant stenosis of the proximal left anterior descending artery, the right coronary artery or the left circumflex artery
* Anginal pain or proven myocardial ischemia due to the coronary stenosis
* Elective percutaneous coronary intervention planned
* Planned direct stenting of the coronary artery

Exclusion Criteria:

* Prior myocardial infarction
* Significant coronary collaterals
* Significant valvular regurgitation (>Sellers II)
* Congestive heart failure
* Pacemaker dependency
* Bundle branch block or significant arrhythmia
* Atrial fibrillation
* Previous coronary bypass grafting
* Impaired kidney function corresponding to a GFR(Glomerular filtration rate) below 60 mL/min.
* Women, who are pregnant or breastfeeding.
* Patient taking part in another clinical study
* Subjects who are committed to an institution and/or penitentiary by judicial or official order.
* Complex coronary lesion requiring balloon angioplasty or rotational atherectomy prior to stenting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
systolic and diastolic function | during 60 seconds ischemia caused by PCI
  Echocardiographic imaging at short intervals of 10 sec during ischemia, which will be induced by elective percutaneous coronary angioplasty with balloon inflation and thus vessel occlusion for 60 sec.

SECONDARY OUTCOMES:
systolic and diastolic function | during 10 minutes, after 1 hour and after 24 hours after PCI
  Echocardiographic imaging of layer specific systolic and diastolic function at intervals of 20 sec during reperfusion up to 10 min after reopening of the vessel as well 1 hour and 24 hours after percutaneous coronary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Hoffmann, Prof.Dr., Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany